CLINICAL TRIAL: NCT02436135
Title: A Phase 1b Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Idelalisib in Subjects Receiving Ruxolitinib as Therapy for Primary, Post-Polycythemia Vera, or Post-Essential Thrombocythemia Myelofibrosis With Progressive or Relapsed Disease
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Idelalisib in Adults Receiving Ruxolitinib as Therapy for Primary, Post-Polycythemia Vera, or Post-Essential Thrombocythemia Myelofibrosis With Progressive or Relapsed Disease
Acronym: Madison
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-397-1245
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — idelalisib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A, Idelalisib + Ruxolitinib (Experimental): Idelalisib 50 mg once daily in participants receiving ruxolitinib.
  Interventions: Drug: Idelalisib; Drug: Ruxolitinib
- Cohort B, Idelalisib + Ruxolitinib (Experimental): Idelalisib 50 mg twice daily in participants receiving ruxolitinib.
  Interventions: Drug: Idelalisib; Drug: Ruxolitinib
- Cohort C, Idelalisib + Ruxolitinib (Experimental): Idelalisib 150 mg once daily in participants receiving ruxolitinib.
  Interventions: Drug: Idelalisib; Drug: Ruxolitinib
- Cohort D, Idelalisib + Ruxolitinib (Experimental): Idelalisib 150 mg twice daily in participants receiving ruxolitinib.
  Interventions: Drug: Idelalisib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib tablets administered orally for 24 weeks
  Other Names: Zydelig®; CAL-101; GS-1101
Drug: Ruxolitinib — Ruxolitinib will be administered per standard of care according to package insert

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, and pharmacokinetics of idelalisib in adults receiving ruxolitinib as therapy for intermediate to high-risk primary myelofibrosis (PMF), post-polycythemia vera, or post-essential thrombocythemia myelofibrosis (post-PV MF or post-ET MF) with progressive or relapsed disease.

This is a dose-escalation study. There will be 4 cohorts (A, B, C, D). Participants will receive an escalating dose or dose frequency of idelalisib based on the safety data of available cohort(s).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals must have been on a stable dose of ruxolitinib for at least 4 weeks prior to study entry
* Individuals with PMF, post-PV MF, or post-ET MF classified as high risk or intermediate risk as defined by the Dynamic International Prognostic Scoring System (DIPSS) for PMF or DIPSS Plus, if cytogenetics are available
* Individuals with PMF, post-PV MF, or post-ET MF who are receiving ruxolitinib and meet 2013 Revised International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) and European Leukemia Net (ELN) response criteria with progressive and relapsed disease, with modifications for progressive disease complete remission (CR), partial remission (PR), or clinical improvement (CI)
* European Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Required screening laboratory values as described in the protocol
* Willing and able to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures, and study restrictions including mandatory prophylaxis for pneumocystis jiroveci pneumonia (PJP)
* Able to understand and willing to sign the informed consent form

Key Exclusion Criteria:

* Individuals on a stable ruxolitinib dose of 5 mg once daily
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing drug-induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver
* Ongoing drug-induced pneumonitis
* Ongoing inflammatory bowel disease
* Ongoing alcohol or drug addiction
* Symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Known hypersensitivity to the study investigational medicinal product (IMP), the metabolites, or formulation excipients
* Unwilling or unable to take oral medication
* Unresolved non-hematologic toxicities from prior therapies that are > Common terminology Criteria for Adverse Events (CTCAE) Grade 1 (with the exception of alopecia [Grade 1 or 2 permitted])
* Pregnant or lactating females
* Cytomegalovirus (CMV): Ongoing infection, treatment, or prophylaxis within the past 28 days

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- United States (2):
  - Stanford Hospital and Clinics, Stanford, California
  - University of Michigan Health System, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 05 June 2015. The last study visit occurred on 20 November 2017.
Pre-assignment Details: 12 participants were screened. Participants were enrolled in Cohorts A and B. After the fourth participant in Cohort B was enrolled, the study was terminated. No additional participants were enrolled.
Groups:
- Cohort A, Idelalisib + Ruxolitinib: Idelalisib tablet 50 mg orally once daily for 24 weeks in participants receiving ruxolitinib as therapy for primary myelofibrosis (PMF), post- polycythemia vera (PV) myelofibrosis (MF), or post-essential thrombocythemia (ET) MF.
- Cohort B, Idelalisib + Ruxolitinib: Idelalisib tablet 50 mg orally twice daily for 24 weeks in participants receiving ruxolitinib as therapy for PMF, post-PV myelofibrosis or post-ET MF.
Period: Overall Study
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Started | 6 | 4
Completed | 0 | 0
Not Completed | 6 | 4
Not completed — Progressive Disease | 3 | 1
Not completed — Investigator Discretion | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Participant | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Cohort A, Idelalisib + Ruxolitinib: Idelalisib tablet 50 mg orally once daily for 24 weeks in participants receiving ruxolitinib as therapy for PMF, post- PV myelofibrosis, or post-ET MF.
- Total: Total of all reporting groups
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10.5) | 69 (6.1) | 65 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 3 | 8
  Others | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Treatment Emergent Adverse Events Within 28 Days of Idelalisib Exposure
Time Frame: First dose date up to 28 days
Population: Full Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants | 100.0 | 75.0

2. Primary Outcome: Percentage of Participants Experiencing Adverse Events Related to Idelalisib Within 28 Days of Idelalisib Exposure
Time Frame: First dose date up to 28 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants | 33.3 | 0

3. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Within 28 Days of Idelalisib Exposure by Worst Grade at Postbaseline
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant. Treatment-emergent laboratory abnormalities were graded per Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 where 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening.
Time Frame: First dose date up to 28 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants
  Anemia (Grade 1) | 0 | 0
  Anemia (Grade 2) | 0 | 0
  Anemia (Grade 3) | 16.7 | 25.0
  Anemia (Grade 4) | 0 | 0
  White blood cell decreased (Grade 1) | 0 | 0
  White blood cell decreased (Grade 2) | 0 | 25.0
  White blood cell decreased (Grade 3) | 0 | 0
  White blood cell decreased (Grade 4) | 0 | 0
  Lymphocyte count decreased (Grade 1) | 0 | 0
  Lymphocyte count decreased (Grade 2) | 33.3 | 0
  Lymphocyte count decreased (Grade 3) | 16.7 | 25.0
  Lymphocyte count decreased (Grade 4) | 0 | 0
  Lymphocyte count increased (Grade 1) | 0 | 0
  Lymphocyte count increased (Grade 2) | 16.7 | 0
  Lymphocyte count increased (Grade 3) | 0 | 0
  Lymphocyte count increased (Grade 4) | 0 | 0
  Neutrophil count decreased (Grade 1) | 0 | 0
  Neutrophil count decreased (Grade 2) | 0 | 25.0
  Neutrophil count decreased (Grade 3) | 0 | 0
  Neutrophil count decreased (Grade 4) | 0 | 0
  Platelet count decreased (Grade 1) | 0 | 25.0
  Platelet count decreased (Grade 2) | 0 | 25.0
  Platelet count decreased (Grade 3) | 16.7 | 0
  Platelet count decreased (Grade 4) | 0 | 0
  Alanine aminotransferase increased (Grade 1) | 16.7 | 25.0
  Alanine aminotransferase increased (Grade 2) | 0 | 0
  Alanine aminotransferase increased (Grade 3) | 0 | 0
  Alanine aminotransferase increased (Grade 4) | 0 | 0
  Hypocalcemia (Grade 1) | 0 | 25.0
  Hypocalcemia (Grade 2) | 0 | 25.0
  Hypocalcemia (Grade 3) | 0 | 0
  Hypocalcemia (Grade 4) | 0 | 0
  Aspartate aminotransferase increased (Grade 1) | 33.3 | 25.0
  Aspartate aminotransferase increased (Grade 2) | 0 | 0
  Aspartate aminotransferase increased (Grade 3) | 0 | 0
  Aspartate aminotransferase increased (Grade 4) | 0 | 0
  Blood bilirubin increased (Grade 1) | 16.7 | 0
  Blood bilirubin increased (Grade 2) | 0 | 0
  Blood bilirubin increased (Grade 3) | 0 | 0
  Blood bilirubin increased (Grade 4) | 0 | 0
  Creatinine increased (Grade 1) | 16.7 | 50.0
  Creatinine increased (Grade 2) | 0 | 0
  Creatinine increased (Grade 3) | 0 | 0
  Creatinine increased (Grade 4) | 0 | 0
  Gamma Glutamyl Transferase Increased (Grade 1) | 16.7 | 0
  Gamma Glutamyl Transferase Increased (Grade 2) | 0 | 25.0
  Gamma Glutamyl Transferase Increased (Grade 3) | 0 | 0
  Gamma Glutamyl Transferase Increased (Grade 4) | 0 | 0
  Hypoglycemia (Grade 1) | 16.7 | 0
  Hypoglycemia (Grade 2) | 0 | 0
  Hypoglycemia (Grade 3) | 0 | 0
  Hypoglycemia (Grade 4) | 0 | 0
  Hypomagnesemia (Grade 1) | 0 | 25.0
  Hypomagnesemia (Grade 2) | 0 | 0
  Hypomagnesemia (Grade 3) | 0 | 0
  Hypomagnesemia (Grade 4) | 0 | 0
  Hyperkalemia (Grade 1) | 0 | 0
  Hyperkalemia (Grade 2) | 16.7 | 0
  Hyperkalemia (Grade 3) | 0 | 0
  Hyperkalemia (Grade 4) | 0 | 0
  Hyperuricemia (Grade 1) | 33.3 | 25.0
  Hyperuricemia (Grade 2) | 0 | 0
  Hyperuricemia (Grade 3) | 0 | 0
  Hyperuricemia (Grade 4) | 16.7 | 0

4. Primary Outcome: Percentage of Participants Who Permanently Discontinued Idelalisib Due to an Adverse Event Within 28 Days of Idelalisib Exposure
Time Frame: First dose date up to 28 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants | 0.0 | 0.0

5. Secondary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events Beyond 28 Days of Idelalisib Exposure
Time Frame: First dose date up to the last dose date (maximum:15.1 months) plus 30 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants Experiencing Adverse Events Related to Idelalisib Beyond 28 Days of Idelalisib Exposure
Time Frame: First dose date up to the last dose date (maximum:15.1 months) plus 30 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants | 50.0 | 25.0

7. Secondary Outcome: Percentage of Participants Experiencing Abnormal Laboratory Abnormalities Beyond 28 Days of Idelalisib Exposure by Worst Grade at Postbaseline
Description: as for outcome 3
Time Frame: First dose date up to the last dose date (maximum:15.1 months) plus 30 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants
  Anemia (Grade 1) | 0 | 0
  Anemia (Grade 2) | 0 | 0
  Anemia (Grade 3) | 33.3 | 25.0
  Anemia (Grade 4) | 0 | 0
  White blood cell decreased (Grade 1) | 16.7 | 0
  White blood cell decreased (Grade 2) | 0 | 25.0
  White blood cell decreased (Grade 3) | 16.7 | 0
  White blood cell decreased (Grade 4) | 0 | 0
  Lymphocyte count decreased (Grade 1) | 0 | 0
  Lymphocyte count decreased (Grade 2) | 0 | 25.0
  Lymphocyte count decreased (Grade 3) | 50.0 | 50.0
  Lymphocyte count decreased (Grade 4) | 16.7 | 0
  Lymphocyte count increased (Grade 1) | 0 | 0
  Lymphocyte count increased (Grade 2) | 33.3 | 25.0
  Lymphocyte count increased (Grade 3) | 0 | 0
  Lymphocyte count increased (Grade 4) | 0 | 0
  Neutrophil count decreased (Grade 1) | 0 | 0
  Neutrophil count decreased (Grade 2) | 0 | 0
  Neutrophil count decreased (Grade 3) | 16.7 | 25.0
  Neutrophil count decreased (Grade 4) | 0 | 0
  Platelet count decreased (Grade 1) | 0 | 25.0
  Platelet count decreased (Grade 2) | 16.7 | 25.0
  Platelet count decreased (Grade 3) | 16.7 | 25.0
  Platelet count decreased (Grade 4) | 0 | 25.0
  Alanine aminotransferase increased (Grade 1) | 16.7 | 25.0
  Alanine aminotransferase increased (Grade 2) | 0 | 25.0
  Alanine aminotransferase increased (Grade 3) | 0 | 25.0
  Alanine aminotransferase increased (Grade 4) | 0 | 0
  Hypocalcemia (Grade 1) | 0 | 25.0
  Hypocalcemia (Grade 2) | 0 | 25.0
  Hypocalcemia (Grade 3) | 0 | 0
  Hypocalcemia (Grade 4) | 0 | 0
  Alkaline phosphatase increased (Grade 1) | 16.7 | 0
  Alkaline phosphatase increased (Grade 2) | 0 | 0
  Alkaline phosphatase increased (Grade 3) | 0 | 0
  Alkaline phosphatase increased (Grade 4) | 0 | 0
  Aspartate aminotransferase increased (Grade 1) | 50.0 | 50.0
  Aspartate aminotransferase increased (Grade 2) | 0 | 25.0
  Aspartate aminotransferase increased (Grade 3) | 0 | 0
  Aspartate aminotransferase increased (Grade 4) | 0 | 0
  Blood bilirubin increased (Grade 1) | 33.3 | 25.0
  Blood bilirubin increased (Grade 2) | 0 | 0
  Blood bilirubin increased (Grade 3) | 0 | 0
  Blood bilirubin increased (Grade 4) | 0 | 0
  Creatinine increased (Grade 1) | 16.7 | 50.0
  Creatinine increased (Grade 2) | 0 | 0
  Creatinine increased (Grade 3) | 0 | 0
  Creatinine increased (Grade 4) | 0 | 0
  Gamma Glutamyl Transferase Increased (Grade 1) | 50.0 | 25.0
  Gamma Glutamyl Transferase Increased (Grade 2) | 0 | 25.0
  Gamma Glutamyl Transferase Increased (Grade 3) | 16.7 | 50.0
  Gamma Glutamyl Transferase Transferase (Grade 4) | 0 | 0
  Hyperglycemia (Grade 1) | 0 | 0
  Hyperglycemia (Grade 2) | 0 | 0
  Hyperglycemia (Grade 3) | 0 | 25.0
  Hyperglycemia (Grade 4) | 0 | 0
  Hypoglycemia (Grade 1) | 16.7 | 0
  Hypoglycemia (Grade 2) | 0 | 0
  Hypoglycemia (Grade 3) | 0 | 0
  Hypoglycemia (Grade 4) | 0 | 0
  Hypomagnesemia (Grade 1) | 0 | 25.0
  Hypomagnesemia (Grade 2) | 0 | 0
  Hypomagnesemia (Grade 3) | 0 | 0
  Hypomagnesemia (Grade 4) | 0 | 0
  Hyperkalemia (Grade 1) | 0 | 25.0
  Hyperkalemia (Grade 2) | 16.7 | 0
  Hyperkalemia (Grade 3) | 0 | 0
  Hyperkalemia (Grade 4) | 0 | 0
  Hypokalemia (Grade 1) | 0 | 25.0
  Hypokalemia (Grade 2) | 0 | 0
  Hypokalemia (Grade 3) | 0 | 0
  Hypokalemia (Grade 4) | 0 | 0
  Hyponatremia (Grade 1) | 0 | 0
  Hyponatremia (Grade 2) | 0 | 0
  Hyponatremia (Grade 3) | 0 | 25.0
  Hyponatremia (Grade 4) | 0 | 0
  Hyperuricemia (Grade 1) | 33.3 | 0
  Hyperuricemia (Grade 2) | 0 | 0
  Hyperuricemia (Grade 3) | 0 | 0
  Hyperuricemia (Grade 4) | 16.7 | 25.0

8. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Idelalisib Due to an Adverse Event Beyond 28 Days of Exposure
Time Frame: First dose date up to the last dose date (maximum:15.1 months) plus 30 days
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
Percentage of participants | 16.7 | 25.0

9. Secondary Outcome: Rate of Overall Response
Description: Rate of overall response as defined by 2013 Revised International Working Group for Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European Leukemia Net (ELN) response criteria.
Time Frame: Start of treatment to end of treatment ( up to 15.1 months)
Population: The study was prematurely terminated due to safety measures. Complete data were not collected for any participant.
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Plasma Concentration of Idelalisib and GS-563117 (Idelalisib Metabolite)
Time Frame: Predose Week 2, 1.5 hour Week 2, and Predose Week 3
Population: The Pharmacokinetic (PK) Analysis Set included all enrolled participants who took at least 1 dose of study drug and have at least 1 nonmissing postdose value reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
Number analyzed (Participants) | 6 | 4
ng/mL
  Idelalisib: Predose Week 2 | 9.95 (6.534) | 106.83 (107.549)
  Idelalisib: 1.5 hour Postdose Week 2 | 835.00 (487.102) | 760.25 (438.644)
  Idelalisib: Predose Week 3 | 6.67 (1.770) | 90.25 (85.374)
  GS-563117: Predose Week 2 | 396.6 (406.95) | 1156.8 (1252.69)
  GS-563117: 1.5 hour Postdose Week 2 | 1051.4 (692.36) | 1405.5 (1228.45)
  GS-563117: Predose Week 3 | 227.9 (212.10) | 988.0 (1018.05)

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date (maximum:15.1 months) plus 30 days
Description: Full Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Cohort A, Idelalisib + Ruxolitinib | Cohort B, Idelalisib + Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Idelalisib + Ruxolitinib (N=6) | Cohort B, Idelalisib + Ruxolitinib (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Idelalisib + Ruxolitinib (N=6) | Cohort B, Idelalisib + Ruxolitinib (N=4)
*Anaemia (Blood and lymphatic system disorders) | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Eructation (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 3 | 0
Influenza like illness (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Serum ferritin increased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT02436135/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT02436135/SAP_001.pdf